CLINICAL TRIAL: NCT04679129
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose Escalation, Single Center Phase I Study to Evaluate Safety, Tolerability and Pharmacokinetics and Pharmacodynamics (Biomarkers) of ASC42 in Healthy Subjects
Brief Title: Study to Evaluate Safety, Tolerability and Pharmacokinetics and Pharmacodynamics of ASC42 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gannex Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASC42-I-CTP-01
Record Dates: First submitted 2020-12-10; First posted 2020-12-22 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Single Ascending Dose-ASC42 (Experimental): ASC42 tablet，Dose 1，Dose 2，Dose 3，Dose 4，and Dose 5, single dose administration
  Interventions: Drug: ASC42
- Multiple Ascending Dose-ASC42 (Experimental): ASC42 tablet, Dose 1，Dose 2，Dose 3，q.d.×14 days
  Interventions: Drug: ASC42
- Single Ascending Dose-Placebo (Placebo Comparator): Placebo tablet，Dose 1，Dose 2，Dose 3，Dose 4，and Dose 5, single dose administration
  Interventions: Drug: Placebo
- Multiple Ascending Dose-Placebo (Placebo Comparator): Placebo tablet，Dose 1，Dose 2，Dose 3，q.d.×14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASC42 — Oral tablets
  Arms: Multiple Ascending Dose-ASC42; Single Ascending Dose-ASC42
Drug: Placebo — Oral tablets
  Arms: Multiple Ascending Dose-Placebo; Single Ascending Dose-Placebo

SUMMARY:
This is a first in human study of single and multiple ascending doses and food effect of ASC42.

This study consists of 8 cohorts and is divided as follows:

Part Ia: Single ascending doses study including cohorts 1 to 5. Part Ib: A cross-over design of cohort 2 to study the food effect on ASC42 PK. Part II: Multiple ascending doses study including cohorts 6 to 8.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy male and female subjects between 18 to 65 years of age.
* Subjects' weight ≥ 50 kg and BMI within the range of 19 - 29 kg/m2.
* Physical examination and vital signs are within normal range or slightly abnormal.

Key Exclusion Criteria:

* History or current liver disease, or liver injuries.
* A positive HBsAg, HCV Ab and/or HIV Ab.
* Platelet count <150,000/mcL
* INR> 1.2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-06-03 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 21 days
  Occurrence of Serious Adverse Event (SAE), Adverse Event (AE) resulting in treatment discontinuation and/or dose reductions, and AE of special interest, from baseline up to 21 days

SECONDARY OUTCOMES:
AUC of ASC42 | On Day 1 to Day 14 after single or multiple doses, respectively. The entire study will last up to 15 days.
  Evaluate the Area under the plasma concentration versus time curve after single and multiple oral doses of ASC42 administered to healthy volunteers.
Cmax of ASC42 | On Day 1 to Day 14 after single or multiple doses, respectively. The entire study will last up to 15 days.
  Evaluate the Peak Plasma Concentration after single and multiple oral doses of ASC42 administered to healthy volunteers.
t1/2 of ASC42 | On Day 1 to Day 14 after single or multiple doses, respectively. The entire study will last up to 15 days.
  Evaluate the Terminal-Phase Half-Life after single and multiple oral doses of ASC42 administered to healthy volunteers.
CL/F of ASC42 | On Day 1 to Day 14 after single or multiple doses, respectively. The entire study will last up to 15 days.
  Evaluate the Apparent Systemic Clearance after single and multiple oral dose of ASC42 administered to healthy volunteers.
Vd/F of ASC42 | On Day 1 to Day 14 after single or multiple doses, respectively. The entire study will last up to 15 days.
  Evaluate the Apparent Volume of Distribution after single and multiple oral dose of ASC42 administered to healthy volunteers.
Tmax of ASC42 | On Day 1 to Day 14 after single or multiple doses, respectively. The entire study will last up to 15 days.
  Evaluate the Time to reach the maximum plasma concentration after single single and multiple oral doses of ASC42 administered to healthy volunteers.
C4 | On Day 1 to Day 14 after single or multiple doses, respectively. The entire study will last up to 15 days.
  Bile acid precuisor:C4 (7αhydroxy-4-cholesten-3-one)
FGF19 | On Day 1 to Day 14 after single or multiple doses, respectively. The entire study will last up to 15 days.
  Bile acid precursor:FGF19 (Fibroblast growth factor 19)

CONTACTS AND LOCATIONS:
Locations (1):
- ICON early Phase Services LLC, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] He H, Wu JJ. Human Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ASC42, a Novel Farnesoid X Receptor Agonist. Drugs R D. 2023 Dec;23(4):453-464. doi: 10.1007/s40268-023-00444-4. Epub 2023 Nov 2. PMID 37919483